CLINICAL TRIAL: NCT01965886
Title: Medial vs Lateral Approach for Total Knee Replacement on Valgus Knee: Prospective and Randomized Clinical Trial
Brief Title: Medial vs Lateral Approach for Total Knee Replacement on Valgus Knee: a Randomized Clinical Trial
Acronym: ValgusKnee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VALGUSKNEE
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2013-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee; arthroplasty; replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medial approach (Active Comparator): Medial parapatellar approach (classic approach)
  Interventions: Procedure: Medial approach
- Keblish approach (Experimental): Lateral parapatellar approach (Keblish approach)
  Interventions: Procedure: Keblish approach

INTERVENTIONS:
Procedure: Medial approach — Total knee replacement performed through a longitudinal incision medial to the patella
  Other Names: medial parapatellar approach; classic approach
  Arms: Medial approach
Procedure: Keblish approach — Total knee replacement performed through a longitudinal incision lateral to the patella
  Other Names: lateral approach; lateral parapatellar approach
  Arms: Keblish approach

SUMMARY:
The most common surgical approach to perform a total knee replacement is called medial parapatellar approach. It's effective and can be applied virtually to all types of knee deformities. The Keblish approach is an alternative approach which uses the lateral side of the patella to enter the joint. Some orthopaedic surgeons consider the latter approach a better option when facing a valgus deformity of the osteoarthritic knee but there is no convincing evidence on the literature supporting one or another approach. The objective of this study is to compare the medial vs lateral approach for total knee replacement on valgus knee.

DETAILED DESCRIPTION:
Total knee replacement is a procedure for the treatment of advanced knee osteoarthritis. The most common surgical approach to perform a total knee replacement is called medial parapatellar approach, or simply medial approach. It's effective and can be applied virtually to all types of knee deformities. The Keblish approach is an alternative approach which uses the lateral side of the patella to enter the joint. It's also called lateral parapatellar approach. Some orthopaedic surgeons consider the latter approach a better option when facing a valgus deformity of the osteoarthritic knee. Theoretically, the Keblish approach can promote better soft tissue balance and patellar tracking, but there is no convincing evidence on the literature supporting one or another approach for a total knee replacement on valgus knee. The objective of this prospective and randomized clinical trial is to compare the medial vs lateral approach for total knee replacement on valgus knee.

ELIGIBILITY:
Inclusion Criteria:

* Severe osteoarthritis (Kellgren & Lawrence grade 4)
* Valgus deformity of the knee
* Read and sign the informed consent form

Exclusion Criteria:

* Severe pain in other joint (VAS>6)
* Comorbidities or any condition that contraindicate the procedure
* Previous arthroplasty on the index knee

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Knee Score | 1 year
  Evaluation of patient's pain and function using the Knee Society questionnaire

SECONDARY OUTCOMES:
WOMAC | 2 years
  Evaluation of patient's symptoms using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
VAS | 2 years
  Evaluation of patient's symptoms using the VAS (Visual Analogic Scale of pain)
Knee alignment | 6 months
  Radiographic analysis of the knee alignment
Hemoglobin | 3 days
  Analysis of patient's hemoglobin to estimate blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro R Zorzi, MsC, Principal Investigator — University of Campinas
Locations (1):
- Hospital de Clínicas da UNICAMP, Campinas, São Paulo, Brazil